CLINICAL TRIAL: NCT07248709
Title: Comparison of High-Intensity Interval Training and Moderate-Intensity Continuous Training on Executive Functions, Cardiorespiratory and Physical Fitness in Older Adults With Mild Cognitive Impairment
Brief Title: Comparison of High-Intensity Interval Training and Moderate-Intensity Continuous Training in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0268 Sadia Khalid
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
Keywords: High-Intensity Interval Training; Moderate-Intensity Continuous Training; Mild Cognitive Impairment; Executive Function; Physical Fitness; Cardiorespiratory Fitness
MeSH Terms: conditions — Cognitive Dysfunction | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The High-Intensity Interval Training Group (HIIT)
  Interventions: Other: High-Intensity Interval Training (HIIT)
- Group B (Experimental): Moderate-Intensity Continuous Training (MICT)
  Interventions: Other: Moderate-Intensity Continuous Training

INTERVENTIONS:
Other: High-Intensity Interval Training (HIIT) — The HIIT group will engage in 28 min of alternating high-intensity and low-intensity exercise, where the high-intensity phase will be at 85-90% of maximum heart rate for 4 min, followed by a 3-min recovery period at 50-60% of maximum heart rate, repeated four times on a treadmill or stationary bicycle. (RPE ~16 on Borg scale) Total duration will be 38 minutes including warm up and cool down period.
  Arms: Group A
Other: Moderate-Intensity Continuous Training — The MICT group's training will consist of continuous aerobic exercise for 28 min at 60-70% of maximum heart rate on a treadmill or stationary bicycle. (RPE ~13 on Borg scale) Total duration will be 38 minutes including warm up and cool down period.
  Arms: Group B

SUMMARY:
This study aims to determine the effects of High-Intensity Interval Training (HIIT) and Moderate-Intensity Continuous Training (MICT) on cognitive and physical fitness in community-dwelling adults diagnosed with Mild Cognitive Impairment (MCI).

A double-blinded randomized clinical trial will be conducted for ten months at Ruhama Welfare Foundation Society Lahore and Kainat Patient Care and Old Age Home, Lahore. The sample size is calculated through G-power and 68 participants will be recruited through the non-probability convenience sampling technique. Those who meet the inclusion criteria will be randomized into two groups through the online randomizer tool. Both experimental groups will undergo an 8-week intervention, consisting of three sessions per week with alternate-day training of 38 minutes. The HIIT group will perform exercise with each session consisting of four 4-minute intervals at 85-95% of their maximum heart rate, with 3-minute active recovery periods, while the MICT group will engage in continuous exercise for 28 minutes at 70-75% of their maximum heart rate. Assessment will be done at baseline, after the 4th week, 8th week, and follow-up at 12th week.

DETAILED DESCRIPTION:
Mild cognitive impairment is a syndrome defined as cognitive decline greater than expected for an individual's age and education level but that does not interfere notably with activities of daily life. Prevalence in population-based epidemiological studies ranges from 3% to 19% in adults older than 65 years. Some people with mild cognitive impairment seem to remain stable or return to normal over time, but more than half progress to dementia within 5 years. Mild cognitive impairment can thus be regarded as a risk state for dementia. The amnestic subtype of mild cognitive impairment has a high risk of progression to Alzheimer's disease, and it could constitute a prodromal stage of this disorder. One of the main causes of disability and dependency in older adults globally, dementia ranks as the seventh most common cause of all disorders. Globally, there were 55 million dementia sufferers in 2021; by 2030, that figure is expected to rise to 78 million, and by 2050, it will reach 139 million. Thankfully, there is a chance that postponing dementia onset by five years could cut its prevalence in half globally. Compared to just 3% of the age-matched group, 46% of people with mild cognitive impairment (MCI), an intermediate stage between normal cognition and dementia, will develop dementia within three years. As a result, MCI is a crucial phase in stopping dementia from getting worse. The multi-cognitive function of subjects with MCI declines.

HIIT can enhance cognitive performance through increased blood flow to the brain, promoting neurogenesis and synaptic plasticity, which are crucial for cognitive tasks. MICT also supports cognitive function. HIIT often produces superior results in a shorter time frame. HIIT involves short bursts of high-intensity exercise followed by rest or low-intensity periods, leading to significant cardiovascular adaptations such as increased VO2 max and improved heart efficiency. MICT, while beneficial, requires longer durations to achieve comparable gains in cardiorespiratory fitness (CRF). Engaging in regular physical exercise has been shown to delay age-related physiological and cognitive decline, reduce the risk of common diseases, and improve the subjective quality of life. Meanwhile, a large proportion of older adults are insufficiently physically active, potentially increasing societal health-related challenges connected to a growing older population. It is, therefore, important to provide both effective and attractive exercise methods adapted for this group. One of the proposed key factors in maximizing exercise effects is to exercise beyond moderate intensities, as in high-intensity interval training (HIIT). Although aerobic moderate-intensity continuous training (MICT) is performed at intensities below the anaerobic threshold, HIIT is broadly defined as short, repeated work intervals at an external intensity close to (80%-100%), or above (>100%) the intensity that elicits maximum oxygen uptake (Vo2 max), with passive or low intensity recovery between intervals.

While exercise is a promising intervention for cognitive health, the comparative efficacy of High-Intensity Interval Training (HIIT) and Moderate-Intensity Continuous Training (MICT) in older adults with MCI remains underexplored. This research seeks to provide useful insights examining the effects of HIIT and MICT on executive functions, cardiorespiratory fitness, and overall physical fitness. HIIT's potential time efficiency and physiological benefits may offer significant advantages over traditional exercise methods. The findings could inform clinical practice, shape public health guidelines, and lead to more effective exercise interventions, ultimately enhancing the quality of life for older adults at risk of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* older adults who had been diagnosed with MCI according to Peterson's criteria [Montreal Cognitive Assessment (MoCA) score <26 for those with 12 years or more of education and <25 for those with less than 12 years of education; activity of daily living scale ≤23; no clinical diagnosis of dementia]
* older adults who are physically normal (the six-item Katz Activities of Daily Living Scale should all be evaluated as "independent")

Exclusion Criteria:

* Participants who have medical problems or co-morbidities that interdict their participation in the study.
* Unable to walk without an assistive device
* Diagnosed with neurodegenerative diseases such as Alzheimer's disease
* Having regular exercise habits (defined as exercise for ≥150 min per week).
* Participating in other ongoing intervention study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Assessment at baseline, after the 4th week, 8th week, and follow-up at 12th week.
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. It has been extensively validated for its reliability and effectiveness in detecting cognitive deficits.

SECONDARY OUTCOMES:
Cognitive Assessment Battery (CAB) | Assessment at baseline, after the 4th week, 8th week, and follow-up at 12th week.
  The CogniFit Cognitive Assessment Battery (CAB) is designed to evaluate cognitive functions, particularly in individuals with mild cognitive impairment (MCI). The CogniFit CAB aims to assess various cognitive skills, including memory, attention, and executive functions, using a computerized format that allows for efficient administration and scoring. The complete CogniFit CAB typically takes about 30-40 minutes to complete.
Trail Making Test | Assessment at baseline, after the 4th week, 8th week, and follow-up at 12th week.
  The Trail Making Test (TMT) is a widely used neuropsychological assessment tool that evaluates cognitive flexibility, executive function, and processing speed. It consists of two parts: TMT-A and TMT-B, each designed to measure different cognitive abilities. TMT-A: This part requires the participant to connect a series of numbered circles in ascending order (1-2-3-4...). It primarily assesses visuoperceptual abilities, such as visual scanning and motor speed. TMT-B: In this part, participants alternate between numbers and letters (1-A-2-B-3-C...), which adds complexity by requiring task-switching and working memory. This portion reflects higher-order executive functions, including cognitive flexibility and the ability to shift attention between tasks.
The Short Physical Performance Battery (SPPB) | Assessment at baseline, after the 4th week, 8th week, and follow-up at 12th week.
  The Short Physical Performance Battery (SPPB) is an objective assessment tool used to evaluate lower extremity functioning and physical performance in older adults including those with mild cognitive impairment (MCI). It consists of three tests: Balance test, Gait speed test and Chair stand test. Each test is scored from 0-4 points. Total SPPB score ranges from 0 (worst performance) to 12 (best performance).
6-Minute Walk Test (6MWT) | Assessment at baseline, after the 4th week, 8th week, and follow-up at 12th week.
  The 6-Minute Walk Test (6MWT) aims to determine how far a person can walk in 6 minutes on a flat, hard surface. The test evaluates the integrated response of multiple bodily systems during exercise, including the respiratory, cardiovascular, and musculoskeletal systems. The person walks back and forth along a measured course, typically 30 meters long. They are instructed to cover as much distance as possible in 6 minutes. Participants can slow down or rest if needed but should resume walking when able.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Khursheed Oldage Home and Nursing Care, Lahore, Punjab Province
  - Ruhama Welfare Foundation Society, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shao Z, Huang J, Feng H, Hu M. Optimizing the physical activity intervention for older adults with mild cognitive impairment: a factorial randomized trial. Front Sports Act Living. 2024 May 7;6:1383325. doi: 10.3389/fspor.2024.1383325. eCollection 2024. PMID 38774280
- [Background] de Lima NS, De Sousa RAL, Amorim FT, Gripp F, Diniz E Magalhaes CO, Henrique Pinto S, Peixoto MFD, Monteiro-Junior RS, Bourbeau K, Cassilhas RC. Moderate-intensity continuous training and high-intensity interval training improve cognition, and BDNF levels of middle-aged overweight men. Metab Brain Dis. 2022 Feb;37(2):463-471. doi: 10.1007/s11011-021-00859-5. Epub 2021 Nov 11. PMID 34762211
- [Background] Tsai CL, Pai MC, Ukropec J, Ukropcova B. The Role of Physical Fitness in the Neurocognitive Performance of Task Switching in Older Persons with Mild Cognitive Impairment. J Alzheimers Dis. 2016 Apr 23;53(1):143-59. doi: 10.3233/JAD-151093. PMID 27128369
- [Background] Martin-Smith R, Cox A, Buchan DS, Baker JS, Grace F, Sculthorpe N. High Intensity Interval Training (HIIT) Improves Cardiorespiratory Fitness (CRF) in Healthy, Overweight and Obese Adolescents: A Systematic Review and Meta-Analysis of Controlled Studies. Int J Environ Res Public Health. 2020 Apr 24;17(8):2955. doi: 10.3390/ijerph17082955. PMID 32344773
- [Background] Wu Q, Niu X, Zhang Y, Song J, Chi A. A Comparative Study of Inhibition Function between High-Intensity Interval Training and Moderate-Intensity Continuous Training in Healthy People: A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2023 Feb 6;20(4):2859. doi: 10.3390/ijerph20042859. PMID 36833556